CLINICAL TRIAL: NCT03940521
Title: Bioclinical Evaluation of 2 Biomarkers of Aviremic HIV-1 in CD4+ T Cells of Adults Undergoing Treatment
Acronym: RESERVIH32
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Institut de Génétique Moléculaire de Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2018-02/PC-01
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-A infected patients
  Interventions: Other: Bioclinical evaluation

INTERVENTIONS:
Other: Bioclinical evaluation — 50-100ml blood extracted for flow cytometry and qPCR

SUMMARY:
The authors hypothesize that there is a correlation between the percentage of CD4+ T cells expressing CD32a and/or X and the quantity of DNA found in peripheral blood mononuclear cells in patients infected with HIV-1. Also, that there is a correlation between expression of CD32a and/or X and proviral load.

ELIGIBILITY:
Inclusion Criteria:

* Patient infected with aviremic HIV-1 (<20 copies of HIV-1 RNA/ml plasma) undergoing antiretroviral treatment for at least 2 years
* Patient has known duration of infection and treatment
* Patient has known pretherapeutic CD4+ T cell count and viremia
* Patient has known CD4+ T cell count, residual viremia and CD4/CD8 ratio for previous 2 years
* Patient weighs at least 56kg
* The patient is not opposed to their inclusion in the study
* The patient must be a member or beneficiary of a health insurance plan
* Patient at least 18 years old

Exclusion Criteria:

* Patient has an acute infection
* The subject has already been included in the study or is in a period of exclusion determined by a previous study
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient is pregnant, parturient or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aviremic HIV-1 undergoing antiretroviral treatment for at least 2 years. Patients will be divided into 3 groups according to pre-therapeutic CD4+ T cell levels:
  * "Low" (n=16): < 200 CD4+ T cells/mm3,
  * "Medium" (n=16): 200 to 500 CD4+ T cells/mm3,
  * "High" (n=16): >500 CD4+ T cells/mm3.
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of CD4+ T cells expressing CD32 alone | Day 0
  %
Percentage of CD4+ T cells expressing X alone | Day 0
  %
Percentage of CD4+ T cells expressing both CD32 and X | Day 0
  %
Quantification of proviral load | Day 0
  Quantitative PCR; number of copies of HIV-1 DNA per million peripheral blood mononuclear cells

SECONDARY OUTCOMES:
Duration of infection prior to treatment | Day 0
  Months
Duration of treatment | Day 0
  Months
Year treatment commenced | Day 0
  Year
Pre-therapeutic CD4 + T cell count | Day 0
  Number of CD4+ T cells/ microL blood
Pre-therapeutic viremia | Day 0
  Number of copies of HIV-1 RNA/ml plasma
Change in CD4+ T cells over previous 2 years | Day 0
  Number of CD4+ T cells/microL blood lost per year
Change in CD4+ T cells prior to treatment | Day 0
  Number of CD4+ T cells/microL blood lost per year
Change in CD4+ T cells during treatment | Day 0
  Number of CD4+ T cells/microL blood lost per year
Viremia at inclusion into the study | Day 0
  Number of copies of HIV-1 RNA/ml plasma
Viremia during the 2 previous years | Day 0
  Number of copies of HIV-1 RNA/ml plasma
Residual immune activation at inclusion into the study | Day 0
  CD4/CD8 ratio
Residual immune activation during the previous 2 years | Day 0
  CD4/CD8 ratio
Nature of current treatment | Day 0
  Family of molecule
Co-infection with hepatitis C virus | Day 0
  Yes/No
Co-infection with hepatitis B virus | Day 0
  Yes/No
Co-infection with Cytomegalovirus | Day 0
  Yes/No
Co-infection with Epstein-Barr virus | Day 0
  Yes/No
Testing for intact proviral DNA | Day 0
  Number of copies/million cells
Circulating viral RNA sequence | Day 0
  RNA sequence

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Corbeau, MD, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No